CLINICAL TRIAL: NCT05466916
Title: Exercise and Diet Intervention opTimized for Gynecologic Cancer Survivors (EDITS Study): Development, Feasibility, and Acceptability
Brief Title: EDITS Pilot Study for Gynecologic Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never initiated and no participants were enrolled.
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Angela Jacqueline Fong, PhD, Instructor of Medicine at Rutgers Cancer Institute of New Jersey, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro2022000863; CINJ 132205 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-07-11; First posted 2022-07-20 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Gynecologic Cancer
Keywords: Gynecologic Cancer; Multiple health behavior change; Optimization; Cancer survivorship; Physical activity; Diet
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Nutrition Assessment; Educational Status

STUDY DESIGN:
Intervention Model Description: In Aims 2 and 3, a single-arm, pre-/post-study design will be used to assess feasibility and acceptability, and preliminary effects of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise and diet education and instruction (Experimental): The intervention will be 12 weeks in duration. The five intervention components (e.g., educational sessions and instructional sessions) will be supervised. Research staff will conduct the intervention. Participants will be instructed to gradually aim for 30 minutes of physical activity for five days per week by Week 12 Participants will also aim for improved healthy dietary practices including > 200 grams/day (g/d) of fruits and vegetables, > 15 g/d of fiber (whole grains and beans), < 250 g/d of sugar-sweetened drinks and lower percent of total kcal from fast foods18 by Week 12. Sessions will be about 35- to 50-minutes in duration and be structured as follows: (a) review of previous session and an opportunity to ask questions (~5 minutes); (b) presentation of content (20- to 30-minutes); (c) opportunity for questions (~5 minutes); and (d) preview of next sessions and research activity reminders (2- to 3-minutes).
  Interventions: Behavioral: Exercise and diet education and instruction

INTERVENTIONS:
Behavioral: Exercise and diet education and instruction — 1:1 or small group sessions consisting of educational materials and exercise instruction.

SUMMARY:
The main goal in this project is to develop and pilot test a 12-week multiple health behavior change (MHBC) intervention for feasibility and acceptability. The pilot study will be guided by Multiphase Optimization Strategy (MOST) framework, which uses highly efficient experiments to systematically test and compare intervention components' or component levels' individual and combined effects. The goal of the MOST framework is to balance effectiveness with affordability, sustainability, and efficiency.

DETAILED DESCRIPTION:
Aim 1: Develop the MHBC intervention with components optimized for gynecologic cancer survivors (GCS). 1a) To develop the intervention components for physical activity and healthy dietary practices, one-on-one interviews will be conducted with stakeholders including GCS (n≈30; until thematic saturation) and gynecologic oncology clinicians (n≈10; until thematic saturation). Clinician is operationalized as any cancer care health professional with direct gynecologic patient contact. Using directed content analysis, it is anticipated that reasons for low uptake in MHBC interventions and gain insight on preferences for intervention components and characteristics such as component delivery (simultaneous vs. sequential), frequency of contact, delivery modality (in-person vs. remote), and support materials (e.g., workbooks and logs) will be identified. The identified factors and preferences will be mapped onto theoretical tenets and taxonomy to develop intervention components. 1b) To refine intervention design and components we will elicit GCS stakeholder input using a cross-sectional study design with an online questionnaire. A questionnaire will be administered to the same 30 GCS from Study 1a to obtain feedback identify intervention preferences.

Aim 2: Determine the feasibility of the MHBC intervention and acceptability of components optimized among GCS. We will evaluate feasibility and acceptability of the 12-week MHBC intervention with 16 GCS. To determine feasibility, the following will be used: number of intervention participants who enroll, those who complete the study, those complete follow-up measures at Week 13, and attendance. Based on previous MHBC interventions with GCS, it is anticipated that 30% will enroll, 85% will complete the intervention, 75% will complete measures at Week 13, and > 70% of the sessions will be attended. To determine acceptability, satisfaction with intervention components at Week 13 will be measured. It is predicted that 86% intervention group will report high satisfaction (cutoff score: > 5 out 7).

Aim 3 (exploratory): Assess the preliminary effects of the intervention on behavioral and cardiometabolic outcomes. The preliminary effects of the intervention on behavioral outcomes including physical activity, healthy dietary practices, HRQOL and cardiometabolic outcomes including weight, waist circumference, body composition (% body fat), and blood pressure will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Only women will be eligible if they meet the following criteria: :

* 18 years old
* A confirmed diagnosis of gynecologic cancer, Stage > I
* Have completed treatment within five years prior to study commencement and hormonal replacement therapy is acceptable
* Are not active, defined as engaging in < 150 minutes of moderate-to-vigorous physical activity per week
* Have a potential unhealthy diet, defined as consuming < 2.5 servings of fruits and vegetables per day, or fast foods more than once per week over the past month
* Are able to converse in and understand English

Exclusion Criteria:

Women will be excluded if they meet any of the following criteria:

* Respiratory, joint, or cardiovascular problems precluding physical activity as per physical activity safety screening questionnaire;
* Metastatic disease
* Planned elective surgery during the duration of the intervention and/or follow-up that would interfere with participation (e.g., reconstructive surgery).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — A confirmed diagnosis of gynecologic cancer, Stage > I
Enrollment: 0 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Participant retention | Baseline
  Participant retention will be tracked through completion of the intervention, assessments, and questionnaires.
Participant retention | Week 13
  Participant retention will be tracked through completion of the intervention, assessments, and questionnaires.
Participant attendance | Baseline
  The research staff will track participant attendance to the intervention sessions.
Participant attendance | Week 13
  The research staff will track participant attendance to the intervention sessions.
Acceptability | Week 13
  Satisfaction will be assessed using Internet Evaluation and Utility Questionnaire

SECONDARY OUTCOMES:
Physical activity (objective) | Baseline and Week 13
  Participants will where an activity tracker to measure minutes of physical activity, intensity, and steps.
Physical activity (self-report) | Baseline and Week 13
  Physical activity intensity and duration will be measured with an adapted version of the Godin Shephard Leisure Time Physical Activity Questionnaire
Healthy Dietary Practices | Baseline and Week 13
  A food diary for 24 hours will be tracked using the NCI's Automated Self-Administered 24 hours tool
Health-related Quality of Life | Baseline and Week 13
  To assess domains of health-related quality of life including Physical health-related domains include General Health, Physical Functioning, Role Physical, and Body Pain. Mental health-related scales include Vitality, Social Functioning, Role Emotional, and Mental Health using the Short Form-12
Exercise Self-efficacy | Baseline and Week 13
  To assess confidence in one's ability to exercise at a moderate intensity three times per week using the adapted Exercise Self-Efficacy Scale
Outcome expectations | Baseline and Week 13
  To assess the expectations about exercising regularly using the Multidimensional Outcome Expectation for Exercise Scale
Facilitators and impediments | Baseline and Week 13
  Open-ended questions asking participants to list any other facilitators and impediments to engagement in the intervention and multiple health behaviors
Blood pressure | Baseline and Week 13
  Systolic and diastolic blood pressure will be measured with an automated cuff.
Height (m) | Baseline and Week 13
  Medical scale with a height ruler.
Height, weight, waist and hip circumference, and body composition | Baseline and Week 13
  Scale, measuring tape, and bioelectric impedance analysis scale
Weight (kg) | Baseline and Week 13
  Scale
Waist and hip circumferences (m) | Baseline and Week 13
  Measuring tape at the smallest and largest portions of the torso.
Body composition | Baseline and Week 13
  Percent of body fat (%) and lean muscle mass )kg) measured using a bioimpedance analysis scale.
6-minute walk test (m) | Baseline and Week 13
  Meters walked in 6-minutes as proxy for cardiovascular fitness.
Chair sit-to-stand (quantity) | Baseline and Week 13
  The total number of times an individual transitions from seated position to a standing position in 30-seconds. Measure of lower body strength
Arm curl test (quantity) | Baseline and Week 13
  Number of times an individual can curl a 5lb weight using their dominant arm in 30-seconds. Measure of upper body strength

CONTACTS AND LOCATIONS:
Overall Officials: Angela J Fong, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers, Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No